CLINICAL TRIAL: NCT04224740
Title: A Phase II Trial of Pembrolizumab Combined With Cisplatin-based Chemotherapy as First-line Systemic Therapy in Advanced Penile Cancer
Brief Title: Pembrolizumab Combined With Cisplatin-based Chemotherapy as First-line Systemic Therapy in Advanced Penile Cancer
Acronym: HERCULES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACOG 0218
Record Dates: First submitted 2020-01-03; First posted 2020-01-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Penile Carcinoma
Keywords: Penile Neoplasms
MeSH Terms: conditions — Penile Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab plus standard of care chemotherapy (Experimental): -Pembrolizumab combined with standard of care therapy
  * Standard of care therapy: ciplastin 70mg/m² IV D1(or carboplatin AUC 5) plus 5-Fluouracil 1000mg/m²/day IV( continuous infusion on Days 1-4) Q3W for 6 cycles
  Interventions: Drug: Pembrolizumab; Drug: Standard of care therapy

INTERVENTIONS:
Drug: Pembrolizumab — Patients will receive pembrolizumab at the dose of 200mg IV Q3W with maximum duration of 2 years (34 cycles-counting the part combined with chemotherapy)
Drug: Standard of care therapy — Ciplastin 70mg/m² IV D1(or carboplatin AUC 5) plus 5-Fluouracil 1000mg/m²/day IV( continuous infusion on Days 1-4) Q3W for 6 cycles
  Other Names: Cisplatin(or Carboplatin), 5-fluouracil

SUMMARY:
This is a phase II clinical trial evaluating activity, safety and patients reported outcomes of first-line pembrolizumab plus cisplatin (or carboplatin) plus 5-FU for patients with advanced penile squamous cell carcinoma.

The primary endpoint is overall responsa rate according to RECIST v1.1 at week 24.

DETAILED DESCRIPTION:
Advanced penile squamous cell carcinoma is associated with dismal survival rates and a major impact on the quality of life. To date, unresectable or metastatic disease is managed by systemic therapy with platinum-based chemotherapy for patients with good performance status. The median PFS and OS on first-line platinum-based chemotherapy vary between 3-4 and 7-15 months, respectively. Chemotherapy induces objective responses in only 20-30% of penile cancer patients with rare complete responses and systemic treatment has not changed for decades. Therefore, this study's rationale is to explore the efficacy and safety of pembrolizumab combined with standard-of-care cisplatin(or carboplatin) plus 5-fluorouracil as part of the first-line therapy. Patients will receive pembrolizumab 200mg IV every three weeks with a maximum duration of 2 years (34 cycles-counting the combination with chemotherapy) in case of no progressive disease or intolerance. The investigators hypothesized that the combination of immunotherapy with standard cytotoxic chemotherapy may improve the overall response rate by RECIST v1.1 in this patient population.

ELIGIBILITY:
INCLUSION

1. Male participants who are at least 18 years of age on the day of signing informed consent will be enrolled in this study.
2. Patients with penile squamous cell carcinoma with either:

   * metastatic disease (de novo or recurrent), or
   * recurrent locally advanced disease not amenable to curative intent therapy (e.g. surgery, radiotherapy, chemoradiotherapy, etc), or
   * anyT N3 M0 or T4 anyN M0 (stage IV - AJCC 8th) not amenable to curative-intent therapy (e.g. surgery, radiotherapy, chemoradiotherapy, etc).
3. Histologically confirmed diagnosis of penile squamous cell carcinoma (PSCC).
4. Patients with advanced or metastatic PSCC without prior treatment or that progressed after 12 months of (neo) adjuvant chemotherapy completion.
5. Participant must agree to use a contraception.
6. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
7. Have measurable disease based on RECIST v1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
8. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.

   Newly obtained biopsies are preferred to archived tissue.
9. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of enrollment.
10. Have adequate organ function (see Table 1). Specimens must be collected within 10 days prior to the start of study treatment.
11. Have a life expectancy of at least 12 weeks.

EXCLUSION

1. Primary tumor arising from urethra.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to enrollment.
4. Has received prior radiotherapy within 3 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has received a live vaccine within 30 days prior to the first dose of study drug.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of non-penile skin or carcinoma in situ that have undergone potentially curative therapy are not excluded.
9. Has known symptomatic uncontrolled CNS metastases and/or carcinomatous meningitis.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a known history of Human Immunodeficiency Virus (HIV).
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection.
16. Has a known history of active TB (Bacillus Tuberculosis).
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is expecting to father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
20. Subjects who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or subject who are MSD employees directly involved in the conduct of the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 24 weeks
  Proportion of patients with partial or complete response by investigator-assessed RECIST v1.1

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 24 months
  Time from enrollment to progression by investigator-assessed RECIST 1.1 or death
Overall survival (OS) | 36 months
  Time from enrollment to death due to any cause.
Clinical Benefit Rate (CBR) | 24 weeks
  Proportion of patients who have complete, partial response or stable disease by investigator-assessed RECIST v1.1
Health Related Quality of Life (QoL) | 24 weeks
  Comparison of initial and final scores of the European Organization for Research and Treatment (EORTC) C30 questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Cotait Maluf, Principal Investigator — Latin American Cooperative Oncology Group
Locations (11):
- Brazil (11):
  - Oncocentro Ceará (Rede D'or), Fortaleza, Ceará
  - ICC - Instituto do Câncer do Ceará, Fortaleza, Ceará
  - Hospital Universitário de Brasília (HUB-UnB), Brasília, Federal District
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - COB - Clínica Oncológica do Brasil, Belém, Pará
  - CPO - Centro de Pesquisa em Oncologia do Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor de Barretos, Barretos, São Paulo
  - INCA - Instituto Nacional de Câncer, Barretos, São Paulo
  - Hospital Amaral Carvalho de Jaú, Jaú, São Paulo
  - ICESP - Instituto do Câncer do Estado de São Paulo, São Paulo
  - BP - A Beneficência Portuguesa de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cotait Maluf F, Trindade K, Preto D, de Almeida Luz M, Medeiros Milhomem Beato P, Assed Bastos D, Holanda Soares JP, Marcondes Lopes V, Werneck de Carvalho LE, Queiroz Borges Muniz D, Racy DJ, de Jesus RG, Rebelatto TF, Werutsky G, Halabi S, Sabino Marques Monteiro F, Poisl Fay A. Pembrolizumab Plus Platinum-Based Chemotherapy for Patients With Advanced Penile Cancer: The Nonrandomized HERCULES (LACOG 0218) Clinical Trial. JAMA Oncol. 2025 Nov 1;11(11):1314-1320. doi: 10.1001/jamaoncol.2025.3266. PMID 40965911